CLINICAL TRIAL: NCT07241403
Title: The Role of Chronic Inflammation in Modulating Targeted Therapy Efficacy and Predicting Treatment Outcomes in Metastatic Colorectal Cancer
Brief Title: Chronic Inflammation, Plasma Proteins Signature, Survival Outcomes and Clinical Response, in Patients Receiving Bevacizumab Combined With Oxaliplatin-based Chemotherapy (Bev/OX) or Bevacizumab Combined With Irinotecan-based Chemotherapy (Bev/IRI)
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Other Study IDs: O-[2025](65)
Record Dates: First submitted 2025-07-25; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Resistance; Bevacizimab; Inflamation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cancer-derived inflammation attenuates the efficacy of adjuvant chemotherapy (CT) in postoperative or metastatic colorectal cancer (mCRC). However, its role in mCRC patients receiving first-line Bevacizumab combined with chemotherapy (Bev/CT) remains unknown. In this prospective observational study, three Bev/CT regimen cohorts (discovery cohort,n=249; Internal validation cohort: n=115; external validation cohort: n=159) and one CT regimen cohort (n=175) were enrolled. Overall survival served as the primary endpoint; clinical response and progression-free survival were secondary endpoints evaluated during follow-up. Investigators used the serum inflammation ratios to evaluate the association between systemic inflammation and clinical outcomes in Bev/CT- and CT-treated mCRC. Combined analysis of 12 cytokines (flow cytometry) and 92 immuno-oncology proteins (Olink) revealed Bev resistance mechanisms and prognosis-predictive biomarkers in Bev/CT treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mCRC;
* Aged over 18 years;
* Must be able to receive the further treatment in the hospital.

Exclusion Criteria:

* More than two types of malignancies;
* Bacterial or virus infection within one month before diagnosis;
* Taken anti-inflammatory drugs or other forms of chemotherapy before their diagnosis;
* participants whose follow-up was interrupted three months ago without reaching any endpoint.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, all enrolled patients received first-line CT or Bev/CT based on the decisions made by both patients and clinicians. The treatment regimens included: (1) oxaliplatin-based CT (FOLFOX/XELOX, OX), (2) irinotecan-based CT (FOLFIRI/ XELIRI, IRI), (3) Bev combined with oxaliplatin-based CT (Bev/OX), and (4) Bev combined with irinotecan-based CT (Bev/IRI). All the patients underwent at least two cycles of Bev/CT until they either withdrew from the disease, experienced disease progression, or encountered intolerable toxic effects.
Sampling Method: Non-Probability Sample
Enrollment: 698 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From January 2018 to December 2024
  OS is the time from initial diagnosis to death, or the last follow-up

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Form January 2018 to December 2024
  PFS is the time from initial diagnosis to disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Nanchang university, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No